CLINICAL TRIAL: NCT00059280
Title: An Open-label, Multicenter, Multinational Study of the Safety, Efficacy, Pharmacokinetics, and Pharmacodynamics of Recombinant Human Acid Alpha-glucosidase Treatment in Patients Less Than 6 Months Old With Infantile-onset Pompe Disease
Brief Title: A Study of the Safety and Efficacy of rhGAA in Patients With Infantile-onset Pompe Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: AGLU01602
Record Dates: First submitted 2003-04-22; First posted 2003-04-23 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2006-07

CONDITIONS: Glycogen Storage Disease Type II
Keywords: Pompe disease; Glycogen storage disease type II; GSD-II; Acid maltase deficiency disease; Glycogenosis 2
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — GAA protein, human

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: Myozyme

INTERVENTIONS:
Biological: Myozyme — 20 mg/kg qow or 40mg/kg qow
  Other Names: Alglucosidase alfa

SUMMARY:
Pompe disease (also known as glycogen storage disease type II, "GSD-II") is caused by a deficiency of a critical enzyme in the body called acid alpha-glucosidase (GAA). Normally, GAA is used by the body's cells to break down glycogen (a stored form of sugar) within specialized structures called lysosomes. In patients with Pompe disease, an excessive amount of glycogen accumulates and is stored in various tissues, especially heart and skeletal muscle, which prevents their normal function. This study is being conducted to evaluate the safety and effectiveness of recombinant human acid alpha-glucosidase (rhGAA) as a potential enzyme replacement therapy for Pompe disease. Patients diagnosed with infantile-onset Pompe disease who are less than or equal to 6 months old will be studied.

ELIGIBILITY:
Inclusion criteria:

* The patient or the patient's legal guardian(s) must provide written informed consent prior to any study-related procedures being performed;
* The patient must have clinical symptoms (documented in his or her medical record) of infantile-onset Pompe disease. In addition, the patient must have: a. an endogenous GAA activity less than 1% of the mean of the normal range as assessed in cultured skin fibroblasts; AND b. cardiomyopathy (LVMI greater than 65 g/m2) by echocardiography;
* The patient must be no older than 26 weeks and 0 days, when he/she receives the first dose of rhGAA;
* The patient and his/her legal guardian(s) must have the ability to comply with the clinical protocol.

Exclusion criteria:

* Symptoms of respiratory insufficiency, including: a. Oxygen saturation less than 90% in room air as measured by pulse oximetry; OR b. venous PCO2 greater than 55 mmHg on room air OR arterial PCO2 greater than 40 mmHg on room air; c. any ventilator use at the time of enrollment;
* Major congenital abnormality;
* Clinically significant organic disease (with the exception of symptoms relating to Pompe disease), including clinically significant cardiovascular, hepatic, pulmonary, neurologic, or renal disease, or other medical condition, serious intercurrent illness, or extenuating circumstance that, in the opinion of the Investigator, would preclude participation in the trial or potentially decrease survival;
* Use of any investigational product within 30 days prior to study enrollment;
* Received enzyme replacement therapy with GAA from any source.

Max Age: 26 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2003-04; Primary Completion 2005-06 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety profile of MZ | 52 weeks
To estimate the proportion of patients treated w/ MZ who were alive and free of ventilator support at 12 months of age; compared to historical cohort | 52 weeks
Determine PK/PD profile of MZ | 52 weeks
Determine effect of different doses of MZ on safety and efficacy | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (8):
- United States (4):
  - University of Florida College of Medicine, Gainesville, Florida
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Utah Medical Center, Salt Lake City, Utah
- Pediatrique Hopital deBrousse, Lyon, France
- Rambam Medical Center, Haifa, Israel
- National Taiwan University Hospital, Taipei, Taiwan
- Royal Manchester Children's Hospital, Manchester, United Kingdom

REFERENCES:
- [Derived] Kishnani PS, Goldenberg PC, DeArmey SL, Heller J, Benjamin D, Young S, Bali D, Smith SA, Li JS, Mandel H, Koeberl D, Rosenberg A, Chen YT. Cross-reactive immunologic material status affects treatment outcomes in Pompe disease infants. Mol Genet Metab. 2010 Jan;99(1):26-33. doi: 10.1016/j.ymgme.2009.08.003. PMID 19775921